CLINICAL TRIAL: NCT01855321
Title: Effects of Treating Vitamin D Deficiency in Poorly Controlled Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 174-2010
Record Dates: First submitted 2013-03-18; First posted 2013-05-16 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Type 2 Diabetes
Keywords: uncontrolled diabetes; vitamin D deficiency
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Vitamin D Deficiency | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Active Comparator): the cholecalciferol capsule with respect to size and shape and 2) the intervention group will take 1 oral capsule of cholecalciferol 50,000 IU (Bio-Tech Pharmacal, Fayetteville, AR USA) once weekly for 8 weeks followed by 50,000 IU once monthly for 4 months.
  Interventions: Drug: Vitamin D
- Placebo (Placebo Comparator): The placebo capsule is to be identical to the cholecalciferol capsule with respect to size and shape and 2) the intervention group will take 1 oral capsule of cholecalciferol 50,000 IU (Bio-Tech Pharmacal, Fayetteville, AR USA) once weekly for 8 weeks followed by 50,000 IU once monthly for 4 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D — The cholecalciferol capsule with respect to size and shape and 2) the intervention group will take 1 oral capsule of cholecalciferol 50,000 IU (Bio-Tech Pharmacal, Fayetteville, AR USA) once weekly for 8 weeks followed by 50,000 IU once monthly for 4 months.
  Other Names: cholecalciferol
  Arms: Vitamin D
Drug: Placebo — The placebo capsule is to be identical to the cholecalciferol capsule with respect to size and shape and 2) the intervention group will take 1 oral capsule of cholecalciferol 50,000 IU (Bio-Tech Pharmacal, Fayetteville, AR USA) once weekly for 8 weeks followed by 50,000 IU once monthly for 4 months.
  Arms: Placebo

SUMMARY:
This pilot study will investigate the effect of Vitamin D supplementation in improving glucose control with patients with poorly controlled diabetes and concurrent Vitamin D deficiency.

DETAILED DESCRIPTION:
Subject will undergo screening procedures, subject will have blood drawn from a vein in your arm to measure subject's Vitamin D level (about 1 tablespoon).If the subject is eligible based on the results of their blood work and the subject agrees to participate in this study, the subject will return to the clinic to begin the study. There will be 4 study visits every 2 months and phone interviews every 2 weeks during the 6 month study. In the beginning (Visit 1) and end of the study (Visit 4), fasting blood samples will be collected for analysis of fasting plasma glucose, %HbAlc (your long-term sugar control over a 3 month period), calcium, insulin, and Vitamin D level. Urine samples will be collected to determine urinary microalbumin-creatinine ratio (early protein loss in the kidneys). Blood pressure will be measured three times with an automatic blood pressure machine. Height and weight will be measured. A medical history questionnaire will be completed by subjects that will include basic demographics, typical dietary intake, smoking and alcohol history, medical history, as well as list of medications and over-the-counter supplements.

At Visit 1 the subject will be randomized (like the toss of a coin) to receive either a sugar pill or a high dose Vitamin D medication, which the subject will take once a week for 8 weeks and then once a month for 4 months. The subject will have a 50:50 chance of receiving one or the other pill. At Visit 2 and Visit 3, the subject will also get blood work to analyze your calcium and Vitamin D level. At each clinic visit, the subject will also have your blood sugar and high blood pressure managed closely by the study investigators, both of who are doctors (one being a primary care doctor and another being an endocrinology/diabetes doctor), according to a standardized preset flowchart.

This means that the doctors in this study will be controlling the subject's blood sugar and blood pressure values closely and may be changing the subject's blood pressure and/or your blood sugar medications during this study depending on what the subject's blood sugar and blood pressure values are. The subject will be instructed not to have their own primary care doctor or diabetes doctor adjust their diabetes or blood pressure as both will be managed closely by the study doctors during the entire 6 month study period. The subject doctors' will be sent a letter notifying of the subject's participation in the study and be instructed not to adjust any of the subject's blood sugar or blood pressure medications during the entire 6 month study as it will be done closely by the study doctors, as clinically indicated. The subject's doctor will be sent letters after each study visit detailing what changes were done, if any, to your blood sugar and blood pressure medication regimen. The subject will be interviewed on the phone every 2 weeks to assess for any medication adverse reactions and treatment compliance.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of type 2 diabetes (per ADA criteria), on antihyperglycemic medications for at least 6 months and
2. HbAlc value of 7.5%-10% 7-12%for at least 3 months prior to screening, and
3. deficiency level of serum 25 (OH) Vitamin D i.e. below20 25 ng/mL at time of screening, but normal serum calcium values of 8.5-10.5mg/dL and
4. on either angiotensin-converting enzyme inhibitor (ACEi) or angiotensin receptor blockade (ARB) antihypertensive medication

Exclusion Criteria:

1. Any subjects with history of end-stage renal disease or frank proteinuria on urinalysis
2. Any subjects with pregnancy at time of screening
3. Any subjects with history of or current hypercalcemia (serum calcium > 10.5 mg/dL) or disease processes with underlying hypercalcemia pathology including hyperparathyroidism, nephrolithiasis, sarcoidosis, lung or bone malignancy
4. Any subjects with diagnosis of Vitamin D deficiency or insufficiency, previously treated or currently treated with any form of prescription doses of either 1,25(OH)2D3 or 25(OH)D3 supplements exceeding 1000 IU/day
5. Any subjects with malabsorption syndromes, nephrotic syndrome, or on medications that activate steroid or xenobiotic receptors which will interfere with absorption of Vitamin D supplements
6. Any subjects with history of serious neurologic or psychiatric disorders that would interfere with the conduct or completion of the study

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Percentage of improvement in Glycemic control after Vitamin D therapy. | 9 months
  We will measure glycemic control as change in %HbAlc and fasting blood glucose after 9 months of Vitamin D therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Lo, MD, Principal Investigator — University of Florida
Locations (1):
- Shands Medical Plaza, Gainesville, Florida, United States